CLINICAL TRIAL: NCT00783016
Title: Effect of Pain Control on the Diagnosis of Acute Appendicitis on the Diagnostic Accuracy of General Surgeon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Kyuseok Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: KSKim
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Appendicitis
Keywords: appendicitis; diagnosis
MeSH Terms: conditions — Appendicitis; Disease | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Morphine (Experimental)
  Interventions: Drug: Morphine
- Placebo (No Intervention)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine

SUMMARY:
The pain control in surgical abdomen has been in debate in masking the correct diagnosis. We would like to investigate the effect of pain control on the diagnostic accuracy of surgeon in suspicious appendicitis patients.

We would give morphine or placebo to the patients suspected of appendicitis randomly and in double-blinded manner, and then surgeons would exam the patient and give the impression for the possibility of the appendicitis(grading 1 to 4).

With this grading, we compare these impression between two groups.

ELIGIBILITY:
Inclusion Criteria:

* the patients suspected of acute appendicitis over 15 years

Exclusion Criteria:

* less than 15 years
* pregnant
* allergic to morphine
* systolic blood pressure<100mmHg
* received pain killer prior to ED visit
* do not consent

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
AUC of ROC of the impression of diagnosis for the appendicitis by surgeon

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Emergency room, Seongnam-si, Gyeonggi-do, South Korea